CLINICAL TRIAL: NCT03738449
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability After Oral Administration of CKD-387 and D484 Under Fed Condition in Healthy Adults
Brief Title: The Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of CKD-387 Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 184BE18014
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * Period 1: D484
  * Period 2: CKD-387
  Interventions: Drug: CKD-387; Drug: D484
- Group 2 (Experimental): * Period 1: CKD-387
  * Period 2: D484
  Interventions: Drug: CKD-387; Drug: D484

INTERVENTIONS:
Drug: CKD-387 — Test drug
Drug: D484 — reference drug

SUMMARY:
The purpose of this clinical trial is to evaluate the pharmacokinetics and safety/tolerability after oral administration of CKD-387 and D484 under fed condition in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 55 years
2. Females must be menopause or surgical infertility
3. Signed informed consent form
4. Other inclusion criteria, as defined in the protocol

Exclusion Criteria:

1. History of clinically significant hepatic, renal, nervous, immune, respiratory, endocrine, hemato-oncology, cardiovascular systemic disease or psychosis disorder
2. Clinical laboratory test values are outside the accepted normal range at Screening

   * aspartate aminotransferase(AST), alanine aminotransferase(ALT) > 1.25 times the upper limit of the normal range
   * Total Bilirubin > 1.5 times the upper limit of the normal range
   * creatine phosphokinase(CPK) > 1.5 times the upper limit of the normal range
   * estimated Glomerular Filtration Rate(eGFR, MDRD* formula) < 60 mL/min/1.73m2 (*MDRD: Modification of Diet in Renal Disease)
   * Positive reaction on following tests: Hepatitis B, Hepatitis C, human immunodeficiency virus(HIV) and syphilis
   * systolic blood pressure(SBP) ≥ 150 mmHg or < 90 mmHg, diastolic blood pressure(DBP) > 100 mmHg or < 50 mmHg
3. Subject who smoke heavily or drink caffeine or alcohol continuously and who cannot discontinue smoking, caffeine or alcohol intake during hospitalization
4. Participated in a clinical trial within 90 days prior to 1st IP dosing
5. Not eligible to participate for the study at the discretion of Investigator
6. Other exclusive inclusion criteria, as defined in the protocol

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of Metformin | 0 hour ~ 48 hour after drug administration
  Cmax of Metformin
Area under the plasma concentration of Metformin-time curve from time zero to time of last measurable concentration | 0 hour ~ 48 hour after drug administration
  AUClast of Metformin

SECONDARY OUTCOMES:
Area under the plasma concentration of Metformin-time curve from time zero to infinity | 0 hour ~ 48 hour after drug administration
  AUCinf of Metformin
Time to reach maximum (peak) plasma concentration of Metformin following drug administration | 0 hour ~ 48 hour after drug administration
  Tmax of Metformin
Half-life of Metformin | 0 hour ~ 48 hour after drug administration
  t1/2 of Metformin
Apparent clearance of Metformin | 0 hour ~ 48 hour after drug administration
  CL/F of Metformin
Apparent volume of distribution of Metformin | 0 hour ~ 48 hour after drug administration
  Vd/F of Metformin

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D. M.D., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea